CLINICAL TRIAL: NCT02745457
Title: The Natural Course and the Effect of Treatment on Body Composition in Children With Inflammatory Bowel Disease
Brief Title: Body Composition in Children With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Head of IBD program, Schneider Children's Medical Center, Israel
Other Study IDs: BodPod IBD
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Growth impairment is commonly seen in children diagnosed with inflammatory bowel diseases (IBD), mainly those with Crohn's disease (CD). There is general consensus in the literature that body composition, composed of fat mass and lean mass is altered in children with IBD compared with controls. Evidence regarding the effect of different therapeutic approaches on body composition in children with IBD is scarce and inconsistent. Furthermore, most studies used anthropometric measures and dual energy X-ray absorptiometry (DEXA) for body composition assessment, while information on the usefulness of air displacement plethysmography (ADP) for this assessment is lacking.

Objectives: To assess body composition in children with IBD by ADP and DEXA at diagnosis and at various intervals during follow up.

Design: A prospective cohort study. Setting: Pediatric gastroenterology institute, Schneider Children's Hospital.

Participants: Children 6 year to 17 years who are diagnosed with either CD or ulcerative colitis (UC).

Main outcome measures: Accuracy of ADP in comparison to DEXA and percentage of fat mass and lean mass at diagnosis and during treatment.

Secondary outcome measures: Correlation of body composition to skin fold, mid arm circumference measurements, BMI, inflammatory markers, gender, disease activity and physical activity.

DETAILED DESCRIPTION:
Children diagnosed with either Crohn's disease (CD) or Ulcerative Colitis (UC) under follow-up at the Pediatric gastroenterology institute, Schneider Children's Hospital, will be enrolled. Patients can be enrolled at diagnosis or at any time point during follow-up. Patients' characteristics will be retrieved from their medical files including demographic details, disease phenotype, anthropometric measures, laboratory evaluation, complication and therapeutic regimens. At enrollment all patients will perform body composition assessment by air displacement plethysmography (ADP) and DEXA (no greater than 7 days between the 2 methods of measurement). At one and two years following initial assessment ADP measurement will be repeated, mid arm circumference and skin fold measurements will be taken and the patient will fill a physical activity questionnaire. Disease activity score (either Pediatric Crohn's Disease Activity Index for CD or Pediatric Ulcerative Colitis Activity Index for UC) will be calculated. Similar evaluation will be performed prior and immediately following exclusive enteral nutrition or corticosteroid courses and prior to any biologic therapy initiation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD
* Age: 6 - 17 years ( inclusive)
* Informed consent

Exclusion Criteria:

* Pregnancy
* Non IBD associated chronic diseases
* Morbid obesity

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children at age 6 year to 17 years diagnosed with IBD
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in body composition accorging to treatment treatment is children with IBD over the course of 2 years | 24 months
  Percentage of fat mass and lean mass at diagnosis and during treatment

SECONDARY OUTCOMES:
To assess the accuracy of ADP in comparison to DEXA based measurement of body composition in children with IBD | 24 months
  To assess the validity of ADP in children with IBD using DEXA as a gold standard for body composition
To evaluate the correlation of body composition to skin fold and mid arm circumference measurements in children with IBD | 24 months
To evaluate the correlation of body composition with BMI | 24 months
To evaluate the correlation of body composition with disease activity | 24 months
To evaluate the correlation of body composition with physical activity | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Schenider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided